CLINICAL TRIAL: NCT05306366
Title: Interventional Open-Label Positron Emission Tomography Study Investigating Blood-Brain-Barrier Penetration and Pharmacokinetic Properties of [11C]-Lu AF90103 in Healthy Young Men
Brief Title: A Brain Imaging PET Study of [11C]-Lu AF90103 in Healthy Adult Male Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: H. Lundbeck A/S (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 19739A
Record Dates: First submitted 2022-03-23; First posted 2022-04-01 (Actual); Last update posted 2022-07-14 (Actual); Status verified 2022-07

CONDITIONS: Healthy Young Men

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- [11C]-Lu AF90103 (Experimental): Participants will receive [11C]-Lu AF90103 via an intravenous bolus injection on Day 1.
  Interventions: Drug: [11C]-Lu AF90103

INTERVENTIONS:
Drug: [11C]-Lu AF90103 — PET ligand administrated as a single intravenous bolus injection

SUMMARY:
The main goals of the study are to assess uptake and distribution of Lu AF90103 in the brain when given at tracer levels (microdose) in healthy young men.

ELIGIBILITY:
Inclusion Criteria:

* The participant has a body mass index (BMI) ≥18.5 and ≤30.0 kilograms (kg)/square meter (m^2) at the Screening Visit.
* The participant is, in the opinion of the investigator, generally healthy based on medical history; a physical examination; vital signs; an electrocardiogram (ECG); and the results of the clinical chemistry, hematology, urinalysis, serology, and other laboratory tests.

Exclusion Criteria:

* The participant has taken disallowed medication <1 week prior to the first dose of study drug or <5 half-lives prior to the Screening Visit for any medication taken.
* The participant has or has had any clinically significant immunological, cardiovascular, respiratory, metabolic, renal, hepatic, gastrointestinal, endocrinological, hematological, dermatological, venereal, neurological, or psychiatric disease or other major disorder.
* The participant has had surgery or trauma with significant blood loss <3 months prior to the first dose of study drug.
* The participant is exposed to significant levels of ionizing radiation at work. Note: Other inclusion and exclusion criteria may apply.

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2022-03-23 (Actual); Primary Completion 2022-06-07 (Actual); Study Completion 2022-06-07 (Actual)

PRIMARY OUTCOMES:
Area Under the Time-Activity Curves for Brain up to 90 Minutes (AUCbrain 0-90 min) | Day 1 (predose and up to 90 minutes postdose)
Area Under the Blood Concentrations Over Time for [11C]-Lu AF90103 and Radioactive Metabolites up to 90 Minutes (AUCblood 0-90 min) | Day 1 (predose and up to 90 minutes postdose)
Area Under the Plasma Concentrations Over Time for [11C]-Lu AF90103 and Radioactive Metabolites up to 90 Minutes (AUCplasma 0-90 min) | Day 1 (predose and up to 90 minutes postdose)
Whole Brain-to-Plasma Ratio Expressed by AUCbrain 0-90 min/AUCplasma 0-90 min | Day 1 (predose and up to 90 minutes postdose)
Total Distribution Volume in the Whole Brain (VT brain) | Day 1 (predose and up to 90 minutes postdose)
Ratio Between the Free Concentrations [11C]-Lu AF90103 in Brain Tissue and Plasma (Kp,uu) | Day 1 (predose and up to 90 minutes postdose)

CONTACTS AND LOCATIONS:
Overall Officials: Email contact via H. Lundbeck A/S, Study Director — H. Lundbeck A/S
Locations (1):
- Karolinska Trial Alliance, Huddinge, Sweden